CLINICAL TRIAL: NCT03060512
Title: A Phase IV, Randomized, Multi-Center, Open-Label, Prospective, Crossover Study to Evaluate Patient Preference of Movantik™ Versus Polyethylene Glycol 3350 for Opioid-Induced Constipation (OIC) Treatment
Brief Title: To Evaluate Patient Preference of Movantik and Polyethylene Glycol 3350 for Opioid Induced Constipation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: QuintilesIMS, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D3820L00017
Record Dates: First submitted 2017-02-13; First posted 2017-02-23 (Actual); Results first posted 2018-07-13 (Actual); Last update posted 2018-07-13 (Actual); Status verified 2018-07

CONDITIONS: Opioid Induced Constipation
Keywords: Opioid Induced constipation,; constipation,; laxative,; bowel movement,; Movantik,; Naloxegol
MeSH Terms: conditions — Opioid-Induced Constipation; Constipation | interventions — polyethylene glycol 3350; naloxegol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Crossover Group 1 (Active Comparator): Crossover Group Movantik to Polyethylene Glycol 3350
  2-period, 2-treatment cross-over model: Subjects will be randomized to Movantik during Treatment period 1 (2 weeks), then crossed over to receive Polyethylene Glycol 3350 for Treatment period 2 (2 weeks) after 1 week washout.
  Interventions: Drug: Polyethylene Glycol 3350; Drug: Movantik
- Crossover Group 2 (Active Comparator): Crossover group Polyethylene Glycol 3350 to Movantik
  2-period, 2-treatment cross-over model: Subjects will be randomized to Polyethylene Glycol 3350 during Treatment period 1 (2 weeks), then crossed over to receive Movantik for Treatment period 2 (2 weeks) after 1 week washout.
  Interventions: Drug: Polyethylene Glycol 3350; Drug: Movantik

INTERVENTIONS:
Drug: Polyethylene Glycol 3350 — Polyethylene Glycol 3350, 17 grams of powder to be dissolved in 4 to 8 ounces of water, juice, soda, coffee or tea to be taken once a day.
  Bisacodyl 5mg, 1-3 tablets may be taken by subject who does not experience a bowel movement within 72 hours.
  Other Names: MiraLAX
Drug: Movantik — Movantik 25 mg, 1 tablet taken once a day on an empty stomach at least 1 hour prior to the first meal of the day or 2 hours after the meal.
  Bisacodyl 5mg, 1-3 tablets may be taken by subject who does not experience a bowel movement within 72 hours.
  Other Names: Naloxegol

SUMMARY:
The purpose of this study is to determine whether patients with opioid induced constipation prefer treatment with naloxegol (Movantik) or with Polyethylene Glycol 3350.

DETAILED DESCRIPTION:
This study is a prospective, randomized, open-label crossover study consisting of a 1-week washout period, a 2-week treatment period, another 1-week washout and a final 2-week treatment period. The study will assess the overall patient preference Movantik versus Polyethylene Glycol 3350 for the treatment of their opioid-induced constipation. This study will also evaluate the reasons for patient preference (only among subjects who indicate a preference), patient global impression of change, and change in bowel function over the treatment periods measured by Bowel Function Index. Patient's bowel movement diary will also be collected during the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between the ages of ≥18 and <85 years
* Self-reported active symptoms of OIC (Opioid Induced Constipation) based on components of the Rome IV criteria at screening. Patients should have at least 2 of the following:

  * <3 SBMs (Spontaneous Bowel Movements) per week
  * Straining >25% of defecations
  * Sensation of incomplete evacuation >25% of defecations
  * Lumpy or hard stools >25% of defecations
  * Sensation of anorectal obstruction/blockage >25% of defecations
* Confirmed OIC by BFI (Bowel Function Index) ≥30
* Stable maintenance opioid regimen consisting of a total daily dose of at least 30 mg of oral morphine, or equivalent of 1 or more other opioid therapies
* Willingness to stop all laxatives and other bowel regimens other than specified rescue medication

Exclusion Criteria:

* Pain related to cancer or has a history of cancer within 5 years
* Current constipation or chronic constipation not caused by or related to use of opioids
* History of rectal evacuation disorders, surgery or procedures that can potentially affect pelvic floor function; requirement of using manual maneuvers to facilitate a bowel movement
* Evidence of significant GI structural abnormalities, acute or chronic GI conditions that could post risk to the patient or confound the study results
* Recent surgery that may affect GI motility or increase risk for bowel obstruction or perforation
* Severe hepatic impairment
* Moderate or severe renal impairment
* Condition that may affect the permeability of blood-brain barrier
* Concomitantly using strong or moderate CYP3A4 inhibitors and strong CYP3A4 inducers
* Any other significant and/or progressive medical, surgical, psychiatric, or mental health condition or any significant laboratory findings that could increase the risk of participation in the study or affect the interpretation of study data as determined by the Investigator

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2017-03-02 (Actual); Primary Completion 2017-08-23 (Actual); Study Completion 2017-08-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Scientific Leadership, Study Director — AstraZeneca
Locations (49):
- United States (49):
  - Research Site, Huntsville, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, Anaheim, California
  - Research Site, Lincoln, California
  - Research Site, Los Gatos, California
  - Research Site, North Hollywood, California
  - Research Site, Orange, California
  - Research Site, San Diego, California
  - Research Site, Westminster, California
  - Research Site, DeLand, Florida
  - Research Site, Fort Myers, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Jupiter, Florida
  - Research Site, Lake City, Florida
  - Research Site, Miami, Florida
  - Research Site, Miami Springs, Florida
  - Research Site, North Miami Beach, Florida
  - Research Site, Ormond Beach, Florida
  - Research Site, Plantation, Florida
  - Research Site, Port Orange, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Decatur, Georgia
  - Research Site, Marietta, Georgia
  - Research Site, Bloomington, Illinois
  - Research Site, Brownsburg, Indiana
  - Research Site, Pikesville, Maryland
  - Research Site, Waltham, Massachusetts
  - Research Site, Troy, Michigan
  - Research Site, Wyoming, Michigan
  - Research Site, Biloxi, Mississippi
  - Research Site, St Louis, Missouri
  - Research Site, Omaha, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, Trenton, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Endwell, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Greensboro, North Carolina
  - Research Site, High Point, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Beavercreek, Ohio
  - Research Site, Edmond, Oklahoma
  - Research Site, Collegeville, Pennsylvania
  - Research Site, Levittown, Pennsylvania
  - Research Site, Greer, South Carolina
  - Research Site, Chattanooga, Tennessee
  - Research Site, Kingsport, Tennessee
  - Research Site, West Jordan, Utah

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Argoff CE, Brennan MJ, Camilleri M, Davies A, Fudin J, Galluzzi KE, Gudin J, Lembo A, Stanos SP, Webster LR. Consensus Recommendations on Initiating Prescription Therapies for Opioid-Induced Constipation. Pain Med. 2015 Dec;16(12):2324-37. doi: 10.1111/pme.12937. Epub 2015 Nov 19. PMID 26582720
- [Result] Bell TJ, Panchal SJ, Miaskowski C, Bolge SC, Milanova T, Williamson R. The prevalence, severity, and impact of opioid-induced bowel dysfunction: results of a US and European Patient Survey (PROBE 1). Pain Med. 2009 Jan;10(1):35-42. doi: 10.1111/j.1526-4637.2008.00495.x. Epub 2008 Aug 18. PMID 18721170
- [Result] Camilleri M, Drossman DA, Becker G, Webster LR, Davies AN, Mawe GM. Emerging treatments in neurogastroenterology: a multidisciplinary working group consensus statement on opioid-induced constipation. Neurogastroenterol Motil. 2014 Oct;26(10):1386-95. doi: 10.1111/nmo.12417. Epub 2014 Aug 28. PMID 25164154
- [Result] Chey WD, Webster L, Sostek M, Lappalainen J, Barker PN, Tack J. Naloxegol for opioid-induced constipation in patients with noncancer pain. N Engl J Med. 2014 Jun 19;370(25):2387-96. doi: 10.1056/NEJMoa1310246. Epub 2014 Jun 4. PMID 24896818
- [Result] Coyne KS, LoCasale RJ, Datto CJ, Sexton CC, Yeomans K, Tack J. Opioid-induced constipation in patients with chronic noncancer pain in the USA, Canada, Germany, and the UK: descriptive analysis of baseline patient-reported outcomes and retrospective chart review. Clinicoecon Outcomes Res. 2014 May 23;6:269-81. doi: 10.2147/CEOR.S61602. eCollection 2014. PMID 24904217
- [Result] Coyne KS, Margolis MK, Yeomans K, King FR, Chavoshi S, Payne KA, LoCasale RJ. Opioid-Induced Constipation Among Patients with Chronic Noncancer Pain in the United States, Canada, Germany, and the United Kingdom: Laxative Use, Response, and Symptom Burden Over Time. Pain Med. 2015 Aug;16(8):1551-65. doi: 10.1111/pme.12724. Epub 2015 Mar 20. PMID 25802051
- [Result] Hurst H, Bolton J. Assessing the clinical significance of change scores recorded on subjective outcome measures. J Manipulative Physiol Ther. 2004 Jan;27(1):26-35. doi: 10.1016/j.jmpt.2003.11.003. PMID 14739871
- [Result] Holzer P. New approaches to the treatment of opioid-induced constipation. Eur Rev Med Pharmacol Sci. 2008 Aug;12 Suppl 1(0 1):119-27. PMID 18924451
- [Result] Johanson JF. Review of the treatment options for chronic constipation. MedGenMed. 2007 May 2;9(2):25. PMID 17955081
- [Result] Kumar L, Barker C, Emmanuel A. Opioid-induced constipation: pathophysiology, clinical consequences, and management. Gastroenterol Res Pract. 2014;2014:141737. doi: 10.1155/2014/141737. Epub 2014 May 5. PMID 24883055
- [Result] McGraw T. Safety of polyethylene glycol 3350 solution in chronic constipation: randomized, placebo-controlled trial. Clin Exp Gastroenterol. 2016 Jul 15;9:173-80. doi: 10.2147/CEG.S111693. eCollection 2016. PMID 27486340
- [Derived] Brenner DM, Hu Y, Datto C, Creanga D, Camilleri M. A Randomized, Multicenter, Prospective, Crossover, Open-Label Study of Factors Associated With Patient Preferences for Naloxegol or PEG 3350 for Opioid-Induced Constipation. Am J Gastroenterol. 2019 Jun;114(6):954-963. doi: 10.14309/ajg.0000000000000229. PMID 31058652
- See also: Movantik_D3820L00017_Protocol_Original-26Jan17_Redacted_PDF-A — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=14622&filename=Movantik_D3820L00017_Protocol_Original-26Jan2017_Redacted_PDF-A.pdf
- See also: Movantik_D3820L00017_SAP_Redacted_15Aug2017_PDF-A — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=14622&filename=Movantik_D3820L00017_SAP_Redacted_15Aug2017_PDF-A.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was performed in 53 sites in the United States. First subject first visit: 2 March 2017. Last subject completed: 23 August 2017. The entire planned duration of study participation was up to 7 weeks.
Pre-assignment Details: 350 subjects were screened and 74 subjects failed to meet the inclusion/exclusion criteria. 276 subjects were randomised to a treatment sequence.
Groups:
- Movantik, Then PEG 3350: Subjects received Movantik 25 milligrams (mg) once daily on an empty stomach at least 1 hour prior to the first meal of the day or 2 hours after the meal for 2 weeks (Treatment Period 1). After a washout period of 1 week, subjects then received Polyethylene Glycol 3350 (PEG 3350) 17 grams (g) of powder dissolved in 4 to 8 ounces of fluid to be taken once daily for 2 weeks (Treatment Period 2).
- PEG 3350, Then Movantik: Subjects received PEG 3350 17 g of powder dissolved in 4 to 8 ounces of fluid to be taken once daily for 2 weeks (Treatment Period 1). After a washout period of 1 week, subjects then received Movantik 25 mg once daily on an empty stomach at least 1 hour prior to the first meal of the day or 2 hours after the meal for 2 weeks (Treatment Period 2).
Period: Overall Study
Arm/Group | Movantik, Then PEG 3350 | PEG 3350, Then Movantik
Started | 137 | 139
Treated With Movantik | 136 | 135
Treated With PEG 3350 | 130 | 138
Completed | 130 | 130
Not Completed | 7 | 9
Not completed — Adverse Event | 4 | 6
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Non-compliance with study medication | 1 | 2

BASELINE CHARACTERISTICS:
Population: The baseline population is the Full Analysis Set (FAS) which consisted of all subjects who satisfied the inclusion and exclusion criteria, received study medication, and attended at least one scheduled visit.
Groups:
- Movantik, Then PEG 3350: Subjects received Movantik 25 mg once daily on an empty stomach at least 1 hour prior to the first meal of the day or 2 hours after the meal for 2 weeks (Treatment Period 1). After a washout period of 1 week, subjects then received PEG 3350 17 g of powder dissolved in 4 to 8 ounces of fluid to be taken once daily for 2 weeks (Treatment Period 2).
- Total: Total of all reporting groups
Arm/Group | Movantik, Then PEG 3350 | PEG 3350, Then Movantik | Total
Number analyzed (Participants) | 132 | 138 | 270
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.9 (9.38) | 56.9 (9.65) | 56.4 (9.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87 | 89 | 176
  Male | 45 | 49 | 94
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 21 | 37
  Not Hispanic or Latino | 115 | 117 | 232
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 31 | 22 | 53
  White | 101 | 113 | 214
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Patient Reported Preference for Movantik or PEG 3350 for Opioid-induced Constipation (OIC) Treatment
Description: The Patient Preference Assessment was conducted at Visit 5 using a 7-point scale in subjects with chronic non-cancer pain. The 3 categories were formed by collapsing the 7-point rating scale to: 1. Prefer Movantik (including Strong preference for Movantik, Moderate preference for Movantik, Slight preference for Movantik), 2. No preference, and 3. Prefer PEG 3350 (including Strong preference for PEG 3350, Moderate preference for PEG 3350, and Slight preference for PEG 3350). The number of subjects in each category is presented for the total number of subjects in the Per-Protocol (PP) Set.
Time Frame: From Visit 2 (Day 1) of Treatment Period 1 to Visit 5 (Day 36) of Treatment Period 2 (end of study).
Population: The PP Set consisted of the subset of the FAS subjects who completed the Patient Preference Assessment at Visit 5 (end of study), and who completed the treatment sequence in the order as specified by the randomised treatment sequence, and were not excluded due to an important protocol deviation.
Measure: Count of Participants; unit: Participants
Groups:
- Total (PP Set): All subjects in the PP Set, including those randomised to both the Movantik/PEG 3350 treatment sequence and the PEG 3350/Movantik treatment sequence.
Arm/Group | Total (PP Set)
Number analyzed (Participants) | 246
Participants
  Prefer Movantik | 124
  Prefer PEG 3350 | 118
  No preference | 4

2. Primary Outcome: Patient Reported Preference for Movantik or PEG 3350 for OIC Treatment by Treatment Sequence
Description: The Patient Preference Assessment was conducted at Visit 5 using a 7-point scale in subjects with chronic non-cancer pain. The following categories were the possible responses: Strong preference for Movantik, Moderate preference for Movantik, Slight preference for Movantik, No preference, Slight preference for PEG 3350, Moderate preference for PEG 3350 and Strong preference for PEG 3350. Prefer Movantik included subjects in the categories Strong preference for Movantik, Moderate preference for Movantik and Slight preference for Movantik. Prefer PEG 3350 included subjects in the categories Strong preference for PEG 3350, Moderate preference for PEG 3350 and Slight preference for PEG 3350. Preference for Period 1 treatment and Preference for Period 2 treatment included subjects who preferred the first and second treatments respectively taken within a given treatment sequence. The number of subjects in each category is presented per treatment sequence for subjects in the PP Set.
Time Frame: From Visit 2 (Day 1) of Treatment Period 1 to Visit 5 (Day 36) of Treatment Period 2 (end of study).
Population: The PP Set consisted of the subset of the FAS subjects who completed the Patient Preference Assessment at Visit 5 (end of study), and who completed the treatment sequence in the order as specified by the randomised treatment sequence, and were not excluded due to an important important protocol deviation.
Measure: Count of Participants; unit: Participants
Arm/Group | Movantik, Then PEG 3350 | PEG 3350, Then Movantik
Number analyzed (Participants) | 125 | 121
Participants
  Strong preference for Movantik | 37 | 38
  Moderate preference for Movantik | 14 | 17
  Slight preference for Movantik | 11 | 7
  No preference | 2 | 2
  Slight preference for PEG 3350 | 9 | 8
  Moderate preference for PEG 3350 | 15 | 23
  Strong preference for PEG 3350 | 37 | 26
  Prefer Movantik | 62 | 62
  Prefer PEG 3350 | 61 | 57
  Preference for Period 1 treatment | 62 | 57
  Preference for Period 2 treatment | 61 | 62
Statistical Analysis 1: Comparison: Movantik, Then PEG 3350 vs PEG 3350, Then Movantik; Assessment of the difference in preference for the two treatments (Prefer Movantik, No Preference, Prefer PEG 3350) in subjects who completed the entire treatment sequence; Test type: Other; p = 0.9239, Prescott's test
Statistical Analysis 2: Comparison: Movantik, Then PEG 3350 vs PEG 3350, Then Movantik; Assessment of the difference between preference for treatment in Period 1, preference for treatment in Period 2, no preference; Test type: Other; p = 0.8874, Prescott's test

3. Secondary Outcome: Patient Reported Influence of Each Medication Characteristic Median Scores That Contributed to Their Overall Preference for Movantik or PEG 3350
Description: In order to assess the reason for patient preference of Movantik or PEG 3350, subjects reported on the influence of 5 medication characteristics using a 4-point rating scale. The following were the scale options: efficacy ('worked better to relieve my OIC'), tolerability ('tolerated better'), convenience ('was more convenient'), works quickly ('worked quickly') and works predictably ('worked predictably'). For each characteristic, influence scores were rated as: 0 = No influence, 1 = Mildly influenced, 2 = Moderately influenced or 3 = Strongly influenced. The scale range for each characteristic was from 0 to 3, and the median score for each characteristic is presented for the overall PP Set according to which treatment was preferred.
  The assessment was only completed by subjects who indicated an overall preference.
Time Frame: From Visit 2 (Day 1) of Treatment Period 1 to Visit 5 (Day 36) of Treatment Period 2 (end of study).
Population: as for outcome 1
Measure: Median (Full Range); unit: Score
Groups:
- Preferred Movantik: Subjects who preferred Movantik for the treatment of OIC had selected Strong preference for Movantik, Moderate preference for Movantik or Slight preference for Movantik during the Patient Preference Assessment at Visit 5.
- Preferred PEG 3350: Subjects who preferred PEG 3350 had selected Strong preference for PEG 3350, Moderate preference for PEG 3350 or Slight preference for PEG 3350 during the Patient Preference Assessment at Visit 5.
Arm/Group | Preferred Movantik | Preferred PEG 3350
Number analyzed (Participants) | 124 | 118
Score
  Worked better to relieve my OIC: number analyzed (Participants) | 123 | 117
  Worked better to relieve my OIC | 2.0 [0 to 3] | 2.0 [0 to 3]
  Tolerated better: number analyzed (Participants) | 123 | 117
  Tolerated better | 3.0 [0 to 3] | 3.0 [0 to 3]
  Was more convenient: number analyzed (Participants) | 123 | 117
  Was more convenient | 3.0 [0 to 3] | 1.0 [0 to 3]
  Worked quickly: number analyzed (Participants) | 123 | 117
  Worked quickly | 2.0 [0 to 3] | 2.0 [0 to 3]
  Worked predictably: number analyzed (Participants) | 123 | 117
  Worked predictably | 2.0 [0 to 3] | 2.0 [0 to 3]

4. Secondary Outcome: Patient Reported Influence of Each Medication Characteristic Individual Category Results That Contributed to Their Overall Preference for Movantik or PEG 3350
Description: In order to assess the reason for patient preference of Movantik or PEG 3350, subjects reported on the influence of 5 medication characteristics using a 4-point rating scale. The following were the scale options: efficacy ('worked better to relieve my OIC'), tolerability ('tolerated better'), convenience ('was more convenient'), works quickly ('worked quickly') and works predictably ('worked predictably'). For each characteristic, influence scores were rated as: 0 = No influence, 1 = Mildly influenced, 2 = Moderately influenced or 3 = Strongly influenced. The scale range for each characteristic was from 0 to 3, and the number of subjects in each characteristic category is presented for the overall PP Set according to which treatment was preferred.
  The assessment was only completed by subjects who indicated an overall preference.
Time Frame: From Visit 2 (Day 1) of Treatment Period 1 to Visit 5 (Day 36) of Treatment Period 2 (end of study).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Preferred Movantik | Preferred PEG 3350
Number analyzed (Participants) | 124 | 118
Participants
  Efficacy: No Influence: number analyzed (Participants) | 123 | 117
  Efficacy: No Influence | 4 | 2
  Efficacy: Mildly Influenced: number analyzed (Participants) | 123 | 117
  Efficacy: Mildly Influenced | 18 | 20
  Efficacy: Moderately Influenced: number analyzed (Participants) | 123 | 117
  Efficacy: Moderately Influenced | 40 | 43
  Efficacy: Strongly Influenced: number analyzed (Participants) | 123 | 117
  Efficacy: Strongly Influenced | 61 | 52
  Tolerability: No Influence: number analyzed (Participants) | 123 | 117
  Tolerability: No Influence | 14 | 15
  Tolerability: Mildly Influenced: number analyzed (Participants) | 123 | 117
  Tolerability: Mildly Influenced | 16 | 11
  Tolerability: Moderately Influenced: number analyzed (Participants) | 123 | 117
  Tolerability: Moderately Influenced | 30 | 32
  Tolerability: Strongly Influenced: number analyzed (Participants) | 123 | 117
  Tolerability: Strongly Influenced | 63 | 59
  Convenience: No Influence: number analyzed (Participants) | 123 | 117
  Convenience: No Influence | 5 | 39
  Convenience: Mildly Influenced: number analyzed (Participants) | 123 | 117
  Convenience: Mildly Influenced | 6 | 26
  Convenience: Moderately Influenced: number analyzed (Participants) | 123 | 117
  Convenience: Moderately Influenced | 26 | 17
  Convenience: Strongly Influenced: number analyzed (Participants) | 123 | 117
  Convenience: Strongly Influenced | 86 | 35
  Works Quickly: No Influence: number analyzed (Participants) | 123 | 117
  Works Quickly: No Influence | 15 | 14
  Works Quickly: Mildly Influenced: number analyzed (Participants) | 123 | 117
  Works Quickly: Mildly Influenced | 25 | 30
  Works Quickly: Moderately Influenced: number analyzed (Participants) | 123 | 117
  Works Quickly: Moderately Influenced | 35 | 41
  Works Quickly: Strongly Influenced: number analyzed (Participants) | 123 | 117
  Works Quickly: Strongly Influenced | 48 | 32
  Works Predictably: No Influence: number analyzed (Participants) | 123 | 117
  Works Predictably: No Influence | 11 | 12
  Works Predictably: Mildly Influenced: number analyzed (Participants) | 123 | 117
  Works Predictably: Mildly Influenced | 21 | 15
  Works Predictably: Moderately Influenced: number analyzed (Participants) | 123 | 117
  Works Predictably: Moderately Influenced | 36 | 48
  Works Predictably: Strongly Influenced: number analyzed (Participants) | 123 | 117
  Works Predictably: Strongly Influenced | 55 | 42

5. Secondary Outcome: Patient Global Impression of Change (PGIC) Questionnaire to Compare the Impact of Movantik and PEG 3350 on OIC Symptoms
Description: PGIC was measured on a 7-point scale at the end of each two-week treatment period to assess the subject's impression of the effectiveness of the treatment received for OIC. The scoring was as follows: 1 = No change (or condition has gotten worse); 2 = Almost the same, hardly any change at all; 3 = A little better, but no noticeable change; 4 = Somewhat better, but the change has not made any real difference; 5 = Moderately better, and a slight but noticeable change; 6 = Better and a definite improvement that has made a real and worthwhile difference; and 7 = A great deal better and a considerable improvement that has made all the difference. The score range is from 1 to 7, with 1 indicating the least improvement and 7 indicating the greatest improvement in OIC symptoms.
  Mean score results are presented for each treatment for Visits 3 and 5.
Time Frame: At Visit 3 (Day 15) of Treatment Period 1 and Visit 5 (Day 36) of Treatment Period 2.
Population: The FAS consisted of all subjects who satisfied inclusion and exclusion criteria, received study medication, and attended at least one scheduled visit. Data is presented for subjects with non-missing PGIC data at the end of at least one of the treatment periods.
Measure: Mean (Standard Deviation); unit: Score
Groups:
- Movantik FAS: The Movantik FAS consisted of all subjects who satisfied the inclusion and exclusion criteria, received Movantik, and attended at least one scheduled visit.
- PEG 3350 FAS: The PEG 3350 FAS consisted of all subjects who satisfied the inclusion and exclusion criteria, received PEG 3350, and attended at least one scheduled visit.
Arm/Group | Movantik FAS | PEG 3350 FAS
Number analyzed (Participants) | 267 | 267
Score | 4.5 (1.83) | 4.5 (1.83)
Statistical Analysis 1: Comparison: Movantik FAS vs PEG 3350 FAS; Analysis of variance (ANOVA) model assessing treatment difference in PGIC at Visits 3 and 5 between Movantik and PEG 3350 treatment. Adjustments were performed for treatment, period and sequence; Test type: Other; Least Squares (LS) Means difference = 0.0, 95% CI 2-sided [-0.3 to 0.3], Standard Error of Mean 0.14

6. Secondary Outcome: PGIC Questionnaire Individual Item Results to Compare the Impact of Movantik and PEG 3350 on OIC Symptoms
Description: PGIC was measured on a 7-point scale at the end of each two-week treatment period to assess the subject's impression of the effectiveness of the treatment received for OIC. The subjects selected one of the following PGIC items as their response: 1 = No change (or condition has gotten worse); 2 = Almost the same, hardly any change at all; 3 = A little better, but no noticeable change; 4 = Somewhat better, but the change has not made any real differences; 5 = Moderately better, and a slight but noticeable change; 6 = Better and a definite improvement that has made a real and worthwhile difference; and 7 = A great deal better and a considerable improvement that has made all the difference. The score range is from 1 to 7, with 1 indicating the least improvement and 7 indicating the greatest improvement in OIC symptoms.
  The number of subjects responding to each PGIC item at Visits 3 and/or 5 is presented for each treatment overall.
Time Frame: At Visit 3 (Day 15) of Treatment Period 1 and Visit 5 (Day 36) of Treatment Period 2.
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Movantik FAS | PEG 3350 FAS
Number analyzed (Participants) | 267 | 267
Participants
  PGIC Item 1: number analyzed (Participants) | 262 | 266
  PGIC Item 1 | 23 | 27
  PGIC Item 2: number analyzed (Participants) | 262 | 266
  PGIC Item 2 | 30 | 27
  PGIC Item 3: number analyzed (Participants) | 262 | 266
  PGIC Item 3 | 21 | 20
  PGIC Item 4: number analyzed (Participants) | 262 | 266
  PGIC Item 4 | 38 | 33
  PGIC Item 5: number analyzed (Participants) | 262 | 266
  PGIC Item 5 | 57 | 66
  PGIC Item 6: number analyzed (Participants) | 262 | 266
  PGIC Item 6 | 61 | 65
  PGIC Item 7: number analyzed (Participants) | 262 | 266
  PGIC Item 7 | 32 | 28

7. Secondary Outcome: Mean Change From Baseline at Visit 3/5 in Bowel Function Index (BFI) Questionnaire Scores to Compare the Impact of Movantik and PEG 3350 on OIC Symptoms
Description: The BFI is a 3-item questionnaire administered by a study clinician to measure constipation from the subject's perspective (ease of defecation, feeling of complete evacuation, and personal judgment of constipation). For each item the subject was asked to rate their response on a scale from 0 to 100, where 0 indicates the best response (easy/no diffculty) and 100 the worst response (severe difficulty). The total BFI score was calculated as the mean of the 3 item scores.
  The mean change from baseline in BFI scores at Visits 3 and/or 5 are presented.
Time Frame: From Baseline (Visit 2, Day 1) to Visit 3 (Day 15) and Visit 5 (Day 36).
Population: The FAS consisted of all subjects who satisfied inclusion and exclusion criteria, received study medication, and attended at least one scheduled visit. Data is presented for subjects with non-missing BFI data at the end of at least one of the two week treatment periods.
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Movantik FAS | PEG 3350 FAS
Number analyzed (Participants) | 267 | 267
Score | -25.0 (31.64) | -26.0 (28.82)
Statistical Analysis 1: Comparison: Movantik FAS vs PEG 3350 FAS; Analysis of Covariance (ANCOVA) model assessing treatment difference in BFI change from baseline at Visits 3/5 between Movantik and PEG 3350. Adjustments were performed for for baseline BFI score, treatment, period and sequence; Test type: Other; LS Means difference = -0.9, 95% CI 2-sided [-4.7 to 3.0], Standard Error of Mean 1.95

ADVERSE EVENTS:
Time Frame: Approximately 5 weeks.
Description: The treatment-emergent safety analysis set included all subjects exposed to at least one dose of either study medication and categorised subjects according to the actual treatment received.
Groups:
- Movantik: The Movantik treatment-emergent safety set included all subjects exposed to at least one dose of Movantik.
- PEG 3350: The PEG 3350 treatment-emergent safety set included all subjects exposed to at least one dose of PEG 3350.
Arm/Group | Movantik | PEG 3350
All-Cause Mortality (participants affected / at risk) | 0/271 | 0/268
Serious Adverse Events (participants affected / at risk) | 3/271 | 1/268
Other Adverse Events (participants affected / at risk) | 66/271 | 46/268
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Movantik (N=271) | PEG 3350 (N=268)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0)
Salmonellosis (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Movantik (N=271) | PEG 3350 (N=268)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Diastolic dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 15 (17) | 6 (6)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 10 (10) | 4 (4)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abnormal faeces (Gastrointestinal disorders) | 0 (0) | 1 (1)
Defaecation urgency (Gastrointestinal disorders) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 10 (10) | 4 (4)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Eructation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 9 (9) | 9 (10)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 5 (5)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)
Drug withdrawal syndrome (General disorders) | 2 (2) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (2) | 0 (0)
Oedema (General disorders) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 1 (1)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood lactic acid increased (Investigations) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 6 (6) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Grief reaction (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1)
Nervousness (Psychiatric disorders) | 1 (1) | 0 (0)
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cold sweat (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Institution and PIs shall be entitled to publish or make presentations related to the Study within 2 years of completion of the Study with Sponsor's prior written consent. PIs shall provide the Sponsor with copies of any materials at least thirty (30) days in advance of publication, submission or presentation.

All such publications or presentations shall be consistent with applicable standards, guidelines and laws, not be false or misleading, and not be made for any commercial purpose.

DOCUMENTS (2):
  • Study Protocol (2017-01-26): https://cdn.clinicaltrials.gov/large-docs/12/NCT03060512/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-15): https://cdn.clinicaltrials.gov/large-docs/12/NCT03060512/SAP_001.pdf